CLINICAL TRIAL: NCT01584245
Title: Evaluation of the Efficacy of an Amino Acid Based Formula in Infants
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enough participants enrolled to provide adequate statistical power
Sponsor: Mead Johnson Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group
Other Study IDs: 6009
Record Dates: First submitted 2012-04-23; First posted 2012-04-24 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Cow's Milk Allergy
MeSH Terms: conditions — Milk Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Amino Acid formula

SUMMARY:
This clinical trial will evaluate the efficacy of an amino acid formula in infants with allergic manifestations.

ELIGIBILITY:
Inclusion Criteria:

* Weight loss within the past 4 weeks
* Infants 1-12 months of age feeding a hypoallergenic formula for at least 2 weeks
* Birth weight greater than or equal to 1500 grams
* Solely enteral fed
* Infants with at least one persistent allergy symptom
* No change in medication within 10 days of beginning the study and no plans for change during the first 10 days of the study
* Signed informed consent

Exclusion Criteria:

* History of underlying condition which, in the Investigator's opinion, could interfere with normal growth, development, or assessment of the participant
* Metabolic disease requiring special attention

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2012-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Weight gain | 12 weeks

SECONDARY OUTCOMES:
Allergic manifestations | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Delphine de Boissieu, M.D., Principal Investigator — Centre médical
Locations (5):
- France (5):
  - Centre médical, Boulogne-Billancourt
  - Hôpital Saint Vincent de Paul, Lille
  - Hôpital Armand Trousseau, Paris
  - Hôpital Necker Enfants Malades, Paris
  - Médecine Infantile 1, Vandoeuvre Lés Nancy

REFERENCES:
- [Derived] Vanderhoof J, Moore N, de Boissieu D. Evaluation of an Amino Acid-Based Formula in Infants Not Responding to Extensively Hydrolyzed Protein Formula. J Pediatr Gastroenterol Nutr. 2016 Nov;63(5):531-533. doi: 10.1097/MPG.0000000000001374. PMID 27526059